CLINICAL TRIAL: NCT01626599
Title: Pilot Study to Evaluate a Baseline Prototype Device Designed to Collect ECG (Electrocardiogram) and Accelerometer Data
Brief Title: Study to Evaluate a New Device Designed to Collect Heart Activity and Body Movement Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Organization: LivaNova (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PG-01
Record Dates: First submitted 2012-06-15; First posted 2012-06-25 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Epilepsy
Keywords: ECG; Accelerometer; Device
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assess product useability (Other): All subjects participate in the same arm. This arm completes the primary objective of product usability.
  Interventions: Device: ProGuardian

INTERVENTIONS:
Device: ProGuardian — The investigational system is composed of a sensor, patch, hub, and caregiver application. The sensor is applied externally during periods of nocturnal sleep for up to 7 nights.
  The investigational system:
  * is not implantable and no surgical procedure is required for a human subject to use the devices;
  * is not for use in supporting or sustaining a human life; and
  * is not of substantial importance in diagnosing, curing, mitigating, or treating disease, or otherwise preventing impairment of human health.
  * Contains skin-contacting materials made of medical grade materials (e.g. sold for use as surgical or wound care) with well-established biocompatibility testing profiles.

SUMMARY:
This study is designed to collect data to support development of a novel product designed to sense changes in heart rate or movement during periods of sleep in people with epilepsy. When a potential seizure is detected, the system sends out an audio-visual notification.

DETAILED DESCRIPTION:
This is a prospective, interventional, un-blinded, non-significant risk, multi-site study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria:

1. Five (5) years of age or older
2. Caregiver capable of understanding and willing to comply with instructions provided in English for proper use of the study device as well as scheduled study visits.
3. Guardian/Parent for subjects less than 18 years or with cognitive limitation that would preclude consent must be willing and able to complete informed consent/and HIPAA authorization.
4. A self-reported diagnosis of epilepsy.
5. Currently taking at least one antiepileptic medication.

Caregivers must meet the following inclusion criteria:

1. Eighteen (18) years of age or older
2. Capable of understanding and willing to comply with instructions provided in english for proper use of the study device as well as scheduled study visits
3. Willing and able to complete informed consent and HIPAA authorization.

Exclusion Criteria:

Subjects are not eligible to be enrolled in the study if they meet any of the following exclusion criteria:

1. Any visible skin disorder, condition, or abnormal skin pigmentation which, in the investigators opinion, would interfere with the ability to wear the patch.
2. History of chronic dermatological, medical, or physical conditions that would, in the investigators opinion, preclude topical application of the test products and/or influence the outcome of the test.
3. Known sensitivity or history of irritation to adhesive tape (Latex) and/or topically applied products
4. An implanted defibrillator and/or pacemakers
5. Severe psychiatric disease that in the investigator's judgment would prevent the patient's successful completion of the study.
6. Pregnant and or nursing women (verified by a urine pregnancy test).
7. Currently participating in another clinical study without sponsor approval.
8. Caregiver that is unable to read instructions in the English language.

Exclusion Criteria for Caregiver:

1. Under 18 years of age
2. Not capable of understanding and willing to comply with instructions provided in English for proper use of the study device as well as scheduled study visits

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Assess product useability | Up to 7 nights/7 days
  This study is designed to collect usability data from the intended use population of people with epilepsy and their caregivers to support development of a novel product designed to capture ECG signals and accelerometer data.

SECONDARY OUTCOMES:
Collect ECG and accelerometer data; device wearability; and evaluate adverse events. | Up to 7 nights/7 days
  Assess ECG and accelerometer data, device adhesion and dermal response

CONTACTS AND LOCATIONS:
Overall Officials: Jason Begnaud, Study Director — Cyberonics, Inc.
Locations (5):
- United States (5):
  - United States, Illinois, Chicago, Illinois
  - United States, North Carolina, Charlotte, North Carolina
  - United States, Texas, Austin, Texas
  - United States, Texas, Houston, Texas
  - United States, Texas, San Antonio, Texas